CLINICAL TRIAL: NCT07195409
Title: Examining the Effectiveness of a Data Coaching Process to Increase Child Physical Activity, Perceived Motor Competence, and Staff Physical Activity Promoting Practices: A Randomized Controlled Trial
Brief Title: Data Coaching Process to Address Staff Physical Activity Promoting Behavior and Child Physical Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Peter Stoepker, Associate Professor of Kinesiology, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-13105; Kansas Department of Health (Other Grant/Funding Number: Kansas Department of Health and Enviornment)
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Physical Activity
Keywords: physical activity; staff behavior; motor competence
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (OST-Coach) (Experimental): Intervention arm (OST-Coach) will receive four data coaching sessions on the data collected at intervention sites. Data will be compiled into a data report and then shared back to the site leaders. Data coaching sessions will follow IDPR principles, first session (investigate), second session (design), third session (practice) and fourth session reflect).
  Interventions: Behavioral: Out of School Time Coach (OST-Coach)
- Control Arm (Standard Practice) (No Intervention): Sites will not receive OST-Coach intervention but will receive data reports.

INTERVENTIONS:
Behavioral: Out of School Time Coach (OST-Coach) — Four data coaching session (investigate, design, practice, reflect) will be conducted over an academic year. Each session will involve: a customized site level data report, goal setting and implementing strategies to address child physical activity, motor competence, and staff physical activity promoting behaviors.
  Arms: Intervention Arm (OST-Coach)

SUMMARY:
The goal of this study is to determine whether a data coaching process called Out of School Time Coach (OST-Coach) can increase child physical activity (PA) behavior, perceived motor competence, and staff PA-promoting practices.

Aim 1: Determine the impact that the OST-Coach intervention has on child PA behavior and perceived motor competence. The investigators hypothesize that integrating a targeted data coaching system will increase the amount of PA children engage in during the OST program and enhance their perceived motor competence compared to sites receiving standard practice.

Aim 2: Assess the impact of the OST-Coach intervention on staff PA-promoting practices. The investigators will measure the effectiveness of the OST-Coach intervention by observing staff behavior and assessing their willingness to integrate evidence-based practices during OST programming. It is hypothesized that OST leaders at intervention sites will implement more PA-promoting practices.

Child physical activity will be measured via systematic observation and a survey assessing perceived motor competence. Staff PA-promoting behaviors will be observed via systematic observation and evaluated through a survey to understand the impact of the data coaching process. The intervention is delivered at the staff level, with feedback provided four times throughout the academic year.

ELIGIBILITY:
Inclusion Criteria:

* All student enrolled in the after-school programs at the elementary level

Exclusion Criteria:

* Not enrolled in the after-school program and not at the elementary level.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Child Physical Activity | Through study completion, 1 year.
  To ensure broader dissemination of this work and make it more feasible for OST-related programs to capture PA data, the investigators will measure child PA through systematic observation. Specifically, they will use the System for Observing Play and Leisure Activity in Youth (SOPLAY), a momentary time sampling technique that systematically observes child PA behavior. During a SOPLAY scan, each child in the activity setting is coded as sedentary, walking, or very active. Additional scans can be conducted for females and males to account for potential group-level gender differences. The validity of SOPLAY has been established through heart rate monitoring and accelerometry-based activity monitors.

SECONDARY OUTCOMES:
Staff Physical Activity Promoting Behavior | Through study completion, 1 year
  A modified version of the System for Observing Staff Promoting Physical Activity and Nutrition (SOPSAN) will be used to capture site leader evidence-based PA promoting practices during OST programming. Scans will begin as soon as children enter the OST site and will last during the duration of designated PA related programming. Target areas will be identified within the OST setting before scans begin and five completed scans will be conducted per target area before moving on to scan another identified area.
Child Percieved Motor Competence | Baseline and end of 1 year
  PlaySelf survey will be implemented at baseline and after the completion of 3 data coaching sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in the study, including baseline characteristics, and outcome measures, will be shared. Supporting documents such as the study protocol and statistical analysis plan will also be available. Data will be accessible beginning 12 months after publication for researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting in June 2025 or after the publication of results and will be available for 6 months.
Access Criteria: Access to de-identified participant data will be granted to qualified researchers in the same field, upon submission of a methodologically sound proposal and approval by the study team. Data must be used only for research purposes, and re-identification of participants is prohibited. The data however is observational and there is no possible way to link to child or staff member participating in study.

REFERENCES:
- [Background] Stoepker P, Biber D, Dauenhauer B, Steel C, Carlson JA. The Integration of a Data Sharing Process to Address Out-of-School Time Physical Activity, Locomotor Skills, and Program Leader Behavior: A Pilot Study. Health Promot Pract. 2025 Jul 10:15248399251348168. doi: 10.1177/15248399251348168. Online ahead of print. PMID 40636958
- [Background] Stoepker P, Dzewaltowski DA. Data Coaching: A Strategy to Address Youth Physical Behavior, Motor Competence, and Out-of-School Time Leader Evidence-Based Practices. J Phys Act Health. 2023 Dec 12;21(3):215-217. doi: 10.1123/jpah.2023-0673. Print 2024 Mar 1. No abstract available. PMID 38086365